CLINICAL TRIAL: NCT07018154
Title: Gender Differences in Musculoskeletal Assessment Methods in Patients With Chronic Mechanical Low Back Pain
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Boles Hanna Boles Melk, Bachlor of Physical Therapy, Cairo University, Cairo, Egypt, Cairo University
Other Study IDs: P.T.REC/012/004982
Record Dates: First submitted 2025-05-31; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Gender Differences; Musculoskeletal Assessment; Chronic; Low Back Pain
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Female patients with chronic nonspecific low back pain (NS-LBP).
  Interventions: Other: Musculoskeletal Assessment
- Group B: Male patients with chronic nonspecific low back pain (NS-LBP).
  Interventions: Other: Musculoskeletal Assessment

INTERVENTIONS:
Other: Musculoskeletal Assessment — Patients underwent a musculoskeletal Assessment.

SUMMARY:
This study is an observational test-retest study designed to investigate the effect of gender on core strength, balance, spinal mobility, and hamstring flexibility in patients with chronic non-specific low back pain (NS-LBP).

DETAILED DESCRIPTION:
Low back pain (LBP) is the primary contributor to years of disability. Individual features (age, physical fitness), psychosocial factors (stress, anxiety, and depression), and occupational factors (hard physical work, bending and twisting motions, and vibration) have all been linked to the development of LBP, which is thought to have a complex etiology.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes will be involved.
* Patients suffer from chronic NS-LBP for more than 3 months.
* Patients' age ranges from 18 to 40 years, and body mass index ranges from 18 to 25 kg/m2.
* Patients with sufficient cognitive abilities that enable them to understand and follow instructions.

Exclusion Criteria:

* History of spinal trauma or fractures.
* Osteoporotic patients.
* Patients using analgesics during the last 3 months.
* Pregnant or lactating females.
* Neurological musculoskeletal diseases that affect the lower back (eg, spondylosis, spondylolisthesis, disc injuries).
* Previous spinal surgery.
* Posture deformities.
* Cauda equina symptoms related to the spine, including changes in bowel and bladder control.
* Signs of severe pathology (eg, malignancy, inflammatory disorders).
* Patients with severe psychiatric disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The current study is an observational test-retest study designed to investigate the effect of gender on core strength, balance, spinal mobility, and hamstring flexibility in patients with chronic nonspecific low back pain (NS-LBP).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Core strength | 6 months post-procedure
  Measurement of core strength was done with the patient in the crooked lying position. Then, the cuff of the device was held under the lower back of the patient, and the patient was instructed to press against this cuff, tuck his abdomen, and hold the contraction.

SECONDARY OUTCOMES:
Balance control | 6 months post-procedure
  Romberg's test was used to assess static balance control. Each patient was tested in a single-leg stance with their eyes open on both a stable surface and then on an unstable surface. For the starting position, each patient stands on their dominant leg (determined by the football kicking test), with the unsupported leg in a neutral hip and 90-degree knee flexion position, and their arms crossed at chest level; the examiner observes this position for 60 seconds. In each test condition (SS and SUS), each patient was asked to maintain the position, and the duration for which they held the position was recorded.
Spinal mobility | 6 months post-procedure
  The Mini-Mental State Examination (MMSE) was used to measure lumbar flexion and extension range of motion. The measurements were taken in a neutral standing position. A line connecting the two posterior superior iliac spines was drawn. Then, two points in the middle of the line and 15 cm above were marked. With lumbar flexion or extension, the distance between the two points was measured and subtracted from the 15 cm distance
Hamstring flexibility | 6 months post-procedure
  To begin the hamstring flexibility test, the patient sits on the floor with both feet straight forward against a box. Both knees were pressed down to the floor. With the palms facing downwards, and the hands side by side, the subject stretched forward four times and held the position of maximum reach on the fourth count. The patient was asked to maintain the position for two counts. The most distant line touched by the fingertips of both hands was noted, and the distance was measured in cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University (Physical therapy), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.